CLINICAL TRIAL: NCT02274038
Title: Serial [18F]Fluorothymidine (FLT)PET/CT as a Biomarker of Therapeutic Response in Pemetrexed Therapy for Non-Small Cell Lung Cancer
Brief Title: Serial [18F]Thymidine (FLT)PET/CT as a Biomarker of Response in Pemetrexed Therapy for Non-Small Cell Lung Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LC130313
Record Dates: First submitted 2014-10-04; First posted 2014-10-24 (Estimated); Results first posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Non-small Cell Lung Cancer; Starting Pemetrexed Based Therapy; Unresectable Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

ARMS (1):
- All patients will be enrolled in a single arm of the study (Experimental): All patients enrolled in the study will receive three 18F-thymidine (FLT) PET/CT scans at the following timepoints: before therapy, on the day of starting pemetrexed therapy (within 24 hours of starting pemetrexed) and at 2-4 weeks of starting pemetrexed therapy.
  Interventions: Drug: Baseline 18F-thymidine (FLT) PET/CT; Drug: Post-therapy 18F-thymidine (FLT) PET/CT to assess for pemetrexed induced tumor FLT "flare"; Drug: Post-therapy 18F-thymidine (FLT) PET/CT to assess for pemetrexed induced changes in tumor proliferation

INTERVENTIONS:
Drug: Baseline 18F-thymidine (FLT) PET/CT — FLT is a fluoro-labelled thymidine analog used as a radiotracer of tumor proliferation in PET/CT imaging. This baseline scan will be used to compare post-therapy FLT-PET/CT in order to assess change in tumor accumulation of FLT.
Drug: Post-therapy 18F-thymidine (FLT) PET/CT to assess for pemetrexed induced tumor FLT "flare" — FLT is a fluoro-labelled thymidine analog used as a radiotracer of tumor proliferation in PET/CT imaging. This scan will be performed on the day of starting pemetrexed therapy (within 24hrs of starting pemetrexed) and used to compare to baseline FLT-PET/CT in order to assess change in tumor accumulation of FLT. The objective is to assess for early pemetrexed induced changes in tumor accumulation of FLT known as FLT "flare".
Drug: Post-therapy 18F-thymidine (FLT) PET/CT to assess for pemetrexed induced changes in tumor proliferation — FLT is a fluoro-labelled thymidine analog used as a radiotracer of tumor proliferation in PET/CT imaging. This scan will be performed 2-4 weeks after starting pemetrexed therapy and used to compare to baseline FLT-PET/CT in order to assess change in tumor accumulation of FLT. The objective is to assess for pemetrexed induced changes in tumor accumulation of FLT as a surrogate measure of tumor proliferation.

SUMMARY:
The investigators will test the hypothesis that positron emission tomography (PET) imaging with the imaging agent 18F-thymidine (FLT) can rapidly assess treatment response in patients with unresectable non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
We will test the hypothesis that positron emission tomography (PET) imaging with the imaging agent 18F-thymidine (FLT) can rapidly assess treatment response in patients with non-small cell lung cancer (NSCLC). In particular, we hypothesize that FLT-PET imaging will offer the potential of rapidly triaging therapy efficacy within hours to days following the start of therapy start by non-invasively monitoring metabolic changes in the tumor, rather than the conventional approach of waiting months for tumors to grow or shrink on computed tomography (CT).

We propose two approaches to evaluate the potential of FLT-PET for assessment of response to therapy in NSCLC. In the first, we will exploit a specific effect (the FLT "flare") induced by pemetrexed, which is first-line chemotherapy for non-squamous NSCLC, to evaluate the utility of FLT-PET to assess successful response to pemetrexed (PEM) therapy within 24 hours. In the second approach, we will utilize FLT as a marker of cell proliferation, as has been done in other cancers, to determine whether chemotherapy has produced a decrease in tumor growth at 2 weeks after starting therapy. Since approximately 70% of patients will fail PEM-based therapy, an imaging technique that could reliably detect PEM efficacy in hours to days rather than months would save valuable time and allow for switch to a more effective therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, at least 18 years of age
2. Histologically confirmed non-small cell lung cancer with at least one site of disease > 1 cm by at least one type of standard imaging (e.g. CT, chest x-ray, MRI)
3. Recommended to start systemic therapy which includes pemetrexed and a platinum-based agent.
4. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.
5. Participants must be willing and able to comply with scheduled visits and imaging procedures in the opinion of the investigator or treating physician.

Exclusion Criteria:

1. Females who are pregnant or breast-feeding at the time of screening will not be eligible for this study. Female participants of child-bearing potential will have a urine pregnancy test at the time of the screening visit.
2. Patients with only a single site of primary lung cancer who have undergone or are recommended to undergo radiation therapy to that site will not be eligible, the inclusion of patients who may be undergoing radiation therapy to ancillary disease sites may be allowed to enter the study at the discretion of the PI if it is not felt to affect the ability to capture FLT information for at least one primary site of disease.
3. Patients who have received chemotherapy within 2 weeks of enrollment will be excluded from the study.
4. Patients who have undergone cancer surgery removing a significant portion of active disease, in the opinion of an investigator, within 2 months prior to study enrollment will be excluded.
5. Inability to tolerate imaging procedures in the opinion of the investigator or treating physician
6. Serious or unstable medical or psychological conditions that, in the opinion of the investigator would compromise the subject's safety or successful participation in the study.
7. Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharyn I Katz, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: none of the enrolled patients were excluded from the study
Groups:
- 18F-thymidine (FLT) PET/CT: All patients enrolled receive three 18F-thymidine (FLT) PET/CT scans at the following timepoints: before therapy, on the day of starting pemetrexed therapy (within 24 hours of starting pemetrexed) and at 2-4 weeks of starting pemetrexed therapy.
  Baseline 18F-thymidine (FLT) PET/CT: FLT is a fluoro-labelled thymidine analog and radiotracer of tumor proliferation in PET/CT imaging. This baseline scan will be used to compare post-therapy FLT-PET/CT to assess change in tumor accumulation of FLT.
  Post-therapy 18F-thymidine (FLT) PET/CT to assess for pemetrexed induced tumor FLT "flare": This scan will be performed on the day of starting pemetrexed therapy (within 24hrs of starting pemetrexed) and used to compare to baseline FLT-PET/CT in order to assess change in tumor accumulation of FLT. The objective is to assess for early pemetrexed induced changes in tumor accumulation of FLT known as FLT "flare".
  Post-therapy 18F-thymidine (FLT) PET/CT to assess for pemetrexed induced changes in tumor proliferation: This scan will be performed 2-4 weeks after starting pemetrexed therapy and used to compare to baseline FLT-PET/CT in order to assess change in tumor accumulation of FLT. The objective is to assess for pemetrexed induced changes in tumor accumulation of FLT as a surrogate measure of tumor proliferation.
Period: Overall Study
Arm/Group | 18F-thymidine (FLT) PET/CT
Started | 3
Completed | 2
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: All patients had adenocarcinoma of the lung
Groups:
- 18F-thymidine (FLT) PET/CT: All patients enrolled in the study will receive three 18F-thymidine (FLT) PET/CT scans at the following timepoints: before therapy, on the day of starting pemetrexed therapy (within 24 hours of starting pemetrexed) and at 2-4 weeks of starting pemetrexed therapy.
  Baseline 18F-thymidine (FLT) PET/CT: FLT is a fluoro-labelled thymidine analog used as a radiotracer of tumor proliferation in PET/CT imaging. This baseline scan will be used to compare post-therapy FLT-PET/CT in order to assess change in tumor accumulation of FLT.
  Post-therapy 18F-thymidine (FLT) PET/CT to assess for pemetrexed induced tumor FLT "flare": This scan will be performed on the day of starting pemetrexed therapy (within 24hrs of starting pemetrexed) and used to compare to baseline FLT-PET/CT in order to assess change in tumor accumulation of FLT. The objective is to assess for early pemetrexed induced changes in tumor accumulation of FLT known as FLT "flare".
  Post-therapy 18F-thymidine (FLT) PET/CT to assess for pemetrexed induced changes in tumor proliferation: This scan will be performed 2-4 weeks after starting pemetrexed therapy and used to compare to baseline FLT-PET/CT in order to assess change in tumor accumulation of FLT. The objective is to assess for pemetrexed induced changes in tumor accumulation of FLT as a surrogate measure of tumor proliferation.
Arm/Group | 18F-thymidine (FLT) PET/CT
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
FLTmax [Mean (Standard Deviation); unit: SUV] — FLTMAX: Maximum SUV (standard uptake value) value on FLT-PET/CT scan
  SUV | 4.2 (2)

OUTCOME MEASURES:

1. Primary Outcome: Baseline 18F-thymidine PET/CT (FLT-PET/CT)
Description: A baseline FLT-PET/CT will be performed prior to starting pemetrexed therapy. This scan will be used to compare to post therapy FLT-PET/CT in order to assess change in tumor accumulation of FLT.
Time Frame: Prior to starting pemetrexed based therapy
Population: based on poor recruitment efforts subjects were unable to be analyzed
Arm/Group | 18F-thymidine (FLT) PET/CT
Number analyzed (Participants) | 0

2. Primary Outcome: Post-therapy 18F-thymidine PET/CT (FLT-PET/CT) to Assess Flare Response
Description: FLT-PET/CT will be performed on the day of starting pemetrexed therapy. This scan will be used to compare to baseline FLT-PET/CT in order to assess change in tumor accumulation of FLT for evidence of an FLT "flare" response to pemetrexed therapy.
Time Frame: On the day that pemetrexed therapy is started
Population: based on poor recruitment efforts subjects were unable to be analyzed
Groups:
- 18F-thymidine (FLT) PET/CT: based on poor recruitment efforts subjects were unable to be analyzed
Arm/Group | 18F-thymidine (FLT) PET/CT
Number analyzed (Participants) | 0

3. Primary Outcome: Post-therapy 18F-thymidine PET/CT (FLT-PET/CT) to Assess Tumor Proliferation Response
Description: FLT-PET/CT will be performed at approximately 2-4 weeks following the start of pemetrexed therapy. This scan will be used to compare to baseline FLT-PET/CT in order to assess change in tumor accumulation of FLT for evidence of a tumor proliferation response to pemetrexed therapy.
Time Frame: Approximately 2-4 weeks following start of pemetrexed therapy.
Population: based on poor recruitment efforts subjects were unable to be analyzed
Arm/Group | 18F-thymidine (FLT) PET/CT
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: Overall survival from enrollment to 12 months from enrollment measured in months
Time Frame: 1 year from study enrollment
Measure: Mean (Standard Deviation); unit: months
Groups:
- 18F-thymidine (FLT) PET/CT: overall survival
Arm/Group | 18F-thymidine (FLT) PET/CT
Number analyzed (Participants) | 3
months | 4.1 (3)

5. Secondary Outcome: Progression-free Survival
Description: based on poor recruitment efforts subjects were unable to be analyzed
Time Frame: Within 1 year from study enrollment
Population: based on poor recruitment efforts subjects were unable to be analyzed
Arm/Group | 18F-thymidine (FLT) PET/CT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 hours following exam
Groups:
- Baseline 18F-thymidine PET/CT (FLT-PET/CT): All patients enrolled in the study will receive three 18F-thymidine (FLT) PET/CT scans at the following timepoints: before therapy, on the day of starting pemetrexed therapy (within 24 hours of starting pemetrexed) and at 2-4 weeks of starting pemetrexed therapy.
  Baseline 18F-thymidine (FLT) PET/CT: This baseline scan will be used to compare post-therapy FLT-PET/CT in order to assess change in tumor accumulation of FLT.
  Post-therapy 18F-thymidine (FLT) PET/CT to assess for pemetrexed induced tumor FLT "flare": This scan will be performed on the day of starting pemetrexed therapy (within 24hrs of starting pemetrexed) and used to compare to baseline FLT-PET/CT in order to assess change in tumor accumulation of FLT. The objective is to assess for early pemetrexed induced changes in tumor accumulation of FLT known as FLT "flare".
  Post-therapy 18F-thymidine (FLT) PET/CT to assess for pemetrexed induced changes in tumor proliferation: This scan will be performed 2-4 weeks after starting pemetrexed therapy and used to compare to baseline FLT-PET/CT in order to assess change in tumor accumulation of FLT. The objective is to assess for pemetrexed induced changes in tumor accumulation of FLT as a surrogate measure of tumor proliferation.
Arm/Group | Baseline 18F-thymidine PET/CT (FLT-PET/CT)
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT02274038/Prot_SAP_000.pdf